CLINICAL TRIAL: NCT05625490
Title: Development and Translation of Generator-Produced PET Tracer for Myocardial Perfusion Imaging
Brief Title: Myocardial Perfusion Imaging Galmydar Rest/Stress
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pamela Woodard, MD, Elizabeth E Mallinckrodt Professor of Radiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202107042-2; R01HL142297 (NIH)
Record Dates: First submitted 2022-11-13; First posted 2022-11-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Perfusion imaging; Pharmacological Stress; Positron Emission Tomography; Myocardial Blood Flow
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients with known or suspected disease and normal controls (no known disease) will both undergo [68Ga]Galmydar PET/CT MPI. Normal controls will also undergo [13N]ammonia PET/CT MPI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Asymptomatic Subjects (Normal Controls) (Experimental): Normal control subjects are asymptomatic, without history of cardiovascular disease or significant cardiovascular risk factors. These participants will receive two [68Ga]Galmydar intravenous administrations, 2 mCi during rest and 4 mCi during stress for the [68Ga]Galmydar PET MPI performed on Imaging Day-1. On Imaging Day-2, asymptomatic subjects will receive two single intravenous administrations each of 10 mCi of [13N]Ammonia during the rest and stress PET MPI. [68Ga]Galmydar and [13N]Ammonia imaging visits will be separated by a minimum of 3 days.
  Interventions: Drug: Ga-68 Galmydar; Drug: 13N-ammonia
- Symptomatic Patients with Normal Clinical SPECT or PET (Experimental): Patients in this group have had a clinical SPECT or PET MPI examination that is normal and do not have an invasive coronary angiography (ICA) referral. Participants will receive one [68Ga]Galmydar intravenous administration, 2 mCi during rest for the [68Ga]Galmydar PET MPI.
  Interventions: Drug: Ga-68 Galmydar
- Symptomatic Patients with Abnormal Clinical SPECT or PET (Experimental): Patients in this group have had a clinical SPECT or PET MPI examination that is positive for ischemia in two myocardial segments and have been referred for invasive coronary angiography (ICA) as part of their routine standard-of-care. Subjects will undergo [68Ga]Galmydar PET/CT prior to any intervention. Participants will receive one [68Ga]Galmydar intravenous administration, 2 mCi during rest.
  Interventions: Drug: Ga-68 Galmydar

INTERVENTIONS:
Drug: Ga-68 Galmydar — Intravenous injections of the PET radiotracer [68Ga]Galmydar.
  Other Names: IND 157468
Drug: 13N-ammonia — Two intravenous injections of PET radiotracer [13N]Ammonia.
  Arms: Asymptomatic Subjects (Normal Controls)

SUMMARY:
A single center, phase 0/1 clinical imaging study designed to assess the role of [68Ga]Galmydar PET/CT imaging in human subjects.

DETAILED DESCRIPTION:
The primary objective of the proposed study is to evaluate the potential of [68Ga]Galmydar PET/CT myocardial perfusion imaging (MPI) for the noninvasive detection of coronary artery disease. The study will evaluate [68Ga]Galmydar PET/CT MPI to semi-quantitatively assess regional myocardial perfusion and quantitatively assess myocardial blood flow (MBF) in patients with suspected or known coronary artery disease (CAD) undergoing clinical SPECT or PET MPI. In addition, perfusion and MBF findings with [68Ga]Galmydar will be compared to the results of coronary morphology or stenosis severity in those patients undergoing invasive coronary angiography (ICA) based on abnormal clinical SPECT or PET MPI. The performance of rest/stress [68Ga]Galmydar PET/CT in comparison to [13N]ammonia PET/CT in normal subjects without cardiovascular disease will be performed as a control. Vital signs, serum chemistries, and serum blood counts will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18-99 years of age and any race;
* Have had a prior clinical SPECT or PET MPI positive for ischemia in two myocardial segments and referred for invasive coronary angiography (ICA) or have had a prior clinical SPECT or PET MPI negative for ischemia or healthy adult normal volunteers who are asymptomatic, without history of cardiovascular disease or significant cardiovascular risk factors;

Exclusion Criteria:

* Inability to receive and sign informed consent;
* Percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 6-months prior to clinical SPECT or PET or in the intervening days between clinical SPECT or PET and research PET examination;
* Participants who have received chemotherapeutic agents within 6 months of enrollment;
* Heart failure (left ventricular ejection fraction ≤ 20%);
* Known non-ischemic cardiomyopathy;
* Inability to undergo pharmacologic stress testing with regadenoson (Lexiscan). Contraindications include:

  * Symptomatic bradycardia or second to third degree atrioventricular (AV) block;
  * Pre-existing obstructive lung disease with active wheezing, i.e., COPD, asthma with active wheezing that precludes the safe administration of the pharmacological stress agent according to the approved label;
  * Uncontrolled and severe hypertension (e.g. systolic blood pressure >200 mmHg, diastolic blood pressure >110 mmHg);
  * Baseline hypotension (e.g. systolic blood pressure < 90 mmHg, diastolic blood pressure <50 mmHg);
* Women who are pregnant or breastfeeding;
* Severe claustrophobia;
* Weight ≥ 500 lbs (weight limit of PET/CT table);
* Administration of any diagnostic or therapeutic radiopharmaceutical, not part of this study, within a period either prior to or after equal to 10 half-lives of the radiopharmaceutical;
* Any condition that in the opinion of the Principal Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with collection of the data such as:

  * Inability to lie still or unable to tolerate a supine position with arms up over the head for up to a 60-minute PET scan due to chronic back/shoulder pain or arthritis as assessed by physical examination and/or medical history;
  * Current or past history of major medical illness, i.e. severe kidney or liver problems;
  * Patients who suffer an intervening clinical event such as worsening angina pectoris or myocardial infarction or whom undergo a myocardial revascularization procedure or have myocardial ischemia at rest;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Semiquantitative assessment of 68Ga-Galmydar PET/CT uptake | Up to 120 minutes post-injection of 68Ga-Galmydar
  Assessment of regional (17segment) myocardial uptake on 5-point scale (0 = normal; 4 = absent tracer uptake) per independent blind readout by 3 expert cardiac PET physicians.

SECONDARY OUTCOMES:
Assessment of myocardial blood flow on 68Ga-Galmydar PET/CT | Up to 120 minutes post-injection of 68Ga-Galmydar
  Assessment of regional (17segment) myocardial blood flow (MBF) at stress and rest perfusion on 68Ga-Galmydar PET/CT.
Change in systolic or diastolic blood pressure. | 6 hours from 68Ga-Galmydar injection
  A 20 mmHg change from baseline in either systolic or diastolic blood pressure.
Change in heart rate. | 6 hours from 68Ga-Galmydar injection
  A 20 BPM change in heart rate from baseline.
Clinically significant change in respiratory rate. | 6 hours from 68Ga-Galmydar injection
  A respiratory rate of < 12 or > 20 breaths/min.
Clinically significant elevation in oral temperature | 6 hours from 68Ga-Galmydar injection
  Oral temperature of >100 degrees F.
Number of patients with new AV Block | 6 hours from 68Ga-Galmydar injection
  A change in EKG showing new AV Block (Type 1 or Type 2), Mobitz 2:1, or QTc ≥ 500ms.
Number of patients with new bradycardia | 6 hours from 68Ga-Galmydar injection
  New heart rate < 40 BPM on EKG.
Clinically significant change in serum chemistries: sodium, potassium, chloride, CO2 | 6 hours from 68Ga-Galmydar injection
  Serum chemistries (sodium, potassium, chloride, CO2) measured in mmol/L. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in serum chemistries: glucose, calcium creatinine, BUN, total bilirubin | 6 hours from 68Ga-Galmydar injection
  Serum chemistries (glucose, calcium creatinine, BUN, total bilirubin), measured in mg/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in serum chemistries: total protein, albumin. | 6 hours from 68Ga-Galmydar injection
  Serum chemistries (total protein, albumin), measured in g/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in serum chemistries: alkaline phosphatase, ALT, AST | 6 hours from 68Ga-Galmydar injection
  Serum chemistries (alkaline phosphatase, ALT, AST), measured in U/L. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in white blood cell count (WBC) | 6 hours from 68Ga-Galmydar injection
  White blood cell count measured in WBC/mm3 blood. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in hemoglobin (Hgb) | 6 hours from 68Ga-Galmydar injection
  Hgb measured in g/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in hematocrit (Hct) | 6 hours from 68Ga-Galmydar injection
  Hct measured in %. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in platelets | 6 hours from 68Ga-Galmydar injection
  Platelets measured in platelets/mm3 blood. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in red blood cell count (RBC) | 6 hours from 68Ga-Galmydar injection
  RBC measured in million/mm3. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Clinically significant change in mean corpuscular volume (MCV) | 6 hours from 68Ga-Galmydar injection
  MCV measured in µm3. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Woodard, M.D, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivapackiam J, Laforest R, Sharma V. 68Ga[Ga]-Galmydar: Biodistribution and radiation dosimetry studies in rodents. Nucl Med Biol. 2018 Apr;59:29-35. doi: 10.1016/j.nucmedbio.2017.11.008. Epub 2017 Dec 1. PMID 29454148